CLINICAL TRIAL: NCT00487526
Title: Clinical Evaluation of the Effect of Duodenal Jejunal Bypass on Type Two Diabetes in Non Obese Adults
Brief Title: Duodenal Jejunal Bypass for Type 2 Diabetes (DJBD)
Acronym: DJBD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ferzli, George S., M.D. F.A.C.S. (Individual)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS07006
Record Dates: First submitted 2007-06-11; First posted 2007-06-18 (Estimated); Last update posted 2007-07-11 (Estimated); Status verified 2007-07

CONDITIONS: Diabetes Mellitus
Keywords: Bypass; Duodenal jejunal; type 2 diabetes; non-obese adults
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: duodenal jejunal bypass

SUMMARY:
Study the effect of Duodenal jejunal bypass on human adults with type 2 diabetes.

DETAILED DESCRIPTION:
Adults non obese ( BMI less than 34 ) will undergo duodenal jejunal bypass. The Outcome measures: Blood Sugar, Insulin,HbA1c, CCK,Gastrin, GIP1and 2, Ghrelin, Cholesterol, Triglycerides,FFA, C-Peptide.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 20-65
* Clinical diagnosis of type 2 diabetes
* Non obese with BMI less than 34.
* Oral agents or insulin to control T2DM.
* Inadequate control of diabetes as defined as HbA1c>/7.5
* Understanding of the mechanisms of action of the treatment

Exclusion Criteria:

* Children with type 1 diabetes
* Obese with BMI over 34
* Coagulopathy
* Liver cirrhosis
* Unable to comply with study requirements, follow-up or give valid consent
* Currently pregnant
* Previous upper abdominal surgery
* Inabilty to tolerate general anesthesia

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-06

PRIMARY OUTCOMES:
control of type 2 diabetes in non obese adults | two years

SECONDARY OUTCOMES:
CCK FFA,Cholesterol,Ghrelin,C-peptide,HbA1c,Gastrin,GIP,Triglycerides,Insulin | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: George S Ferzli, MD F.A.C.S, Principal Investigator — SUNY Downstate
Locations (1):
- Center for Advance Medicine Abel Gonzalez, Santo Domingo, Dominican Republic